CLINICAL TRIAL: NCT00040391
Title: A Phase II, Randomized, Open-label, Controlled, Dose-elevation, Multicenter Trial of an Investigational Drug for the Prevention of Diarrhea Associated With Irinotecan/5FU/Leucovorin Chemotherapy in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: A Trial of an Investigational Drug for the Prevention of Diarrhea Associated With Irinotecan/5FU/Leucovorin Chemotherapy in Previously Untreated Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 440E-ONC-0020-315
Record Dates: First submitted 2002-06-26; First posted 2002-06-27 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Neoplasms; Diarrhea
Keywords: Pharmacia
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea | interventions — Drugs, Investigational; Irinotecan; Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: Investigational drug
Drug: Irinotecan
Drug: 5-fluorouracil
Drug: Leucovorin

SUMMARY:
The study will combine a new investigational drug with standard anti-cancer drugs for the treatment of advanced colorectal cancer. The standard and approved treatment for colorectal cancer is to undergo chemotherapy with a combination of irinotecan (also known as CPT-11, Camptosar), 5-fluorouracil (also known as 5-FU), and leucovorin (also known as LV). This is known as the triple therapy. One of the major side effects of CPT-11/5-FU/LV chemotherapy treatment is diarrhea. The purpose of this research study is to see whether adding this investigational drug to the standard treatment for advanced colorectal cancer can reduce the amount of diarrhea a patient experiences. This study will also determine if adding the investigational drug to triple therapy has a positive effect on tumors.

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria:

* Age 18 years or older
* Diagnosis of colorectal cancer or adenocarcinoma of the appendix
* A tumor mass that can be measured
* Resolution of all toxic effects of any radiotherapy or surgical procedures to NCI CTC grade less than or equal to 1
* Willingness and ability to comply with scheduled visits, treatment plan, and laboratory tests, and other study procedures

Exclusion Criteria:

* Women that are pregnant or lactating
* Prior treatment with Irinotecan
* Partial or complete bowel obstruction, known chronic malabsorption, or total colectomy or other major abdominal surgery that might result in substantial alteration in transit or absorption of oral medication
* Administration of the last dose of any previous adjuvant therapy for colorectal cancer within 6 months previous to randomization
* Current enrollment in another clinical trial
* Administration of any prior systemic anticancer therapy for metastatic colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Research Center, Little Rock, Arkansas
  - Research Center, Anaheim, California
  - Research Center, Concord, California
  - Research Center, Gilroy, California
  - Research Center, Los Angeles, California
  - Research Center, Jacksonville, Florida
  - Research Center, New Port Richey, Florida
  - Research Center, New Orleans, Louisiana
  - Research Center, Scarborough, Maine
  - Research Center, Pittsfield, Massachusetts
  - Research Center, East Lansing, Michigan
  - Research Center, Saint Joseph, Michigan
  - Research Center, Minneapolis, Minnesota
  - Research Center, Saint Joseph, Missouri
  - Research Center, Las Vegas, Nevada
  - Research Center, East Setauket, New York
  - Research Center, Northport, New York
  - Research Center, Burlington, North Carolina
  - Research Center, Greenville, North Carolina
  - Research Center, Zanesville, Ohio
  - Research Center, Lancaster, Pennsylvania
  - Research Center, Philadelphia, Pennsylvania
  - Research Center, Charleston, South Carolina
  - Research Center, Germantown, Tennessee
  - Research Center, Dallas, Texas
  - Research Center, Madison, Wisconsin
  - Research Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Pan CX, Loehrer P, Seitz D, Helft P, Juliar B, Ansari R, Pletcher W, Vinson J, Cheng L, Sweeney C. A phase II trial of irinotecan, 5-fluorouracil and leucovorin combined with celecoxib and glutamine as first-line therapy for advanced colorectal cancer. Oncology. 2005;69(1):63-70. doi: 10.1159/000087302. Epub 2005 Aug 2. PMID 16088234